CLINICAL TRIAL: NCT06139835
Title: a Proof of Principle in Vivo Study to Evaluate the Anti-Calculus and Safety Profile of a Novel Enzyme Formulation
Brief Title: Testing if Tartarase Can Remove Dental Tartar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontis Biologics, Inc. (Industry)
Collaborators: Salus Research, Inc., 1220 Medical Park Dr. A, Fort Wayne ID 46825 (Unknown); Reinhard Schuller Consulting, 37 Poplar Heights Dr., Toronto, Ontario M9A 5A1 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB2022-01
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Calculus
Keywords: gingivitis; dentifrice; plaque
MeSH Terms: conditions — Dental Calculus; Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Comparison of the change in calculus abundance of two treatment groups, using the same dentifrice with two different methods of application with a control group using a popular standard dentifrice.
Who Masked: Care Provider
Masking Description: The group of study subjects, selected from the study site's database were randomized by the statistician into three different treatment groups. The personnel performing the measurements were blinded as to which group the study subjects we in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Individuals randomly assigned to the control arm where they brushed their teeth with a popular toothpaste (crest) in the morning and before bed. This routine was repeated daily for 4 weeks.
  Interventions: Biological: Tartarase
- Tartarase brushing (Experimental): In the morning, this group brushed with Tartarase for 30 seconds, spit, but did not rinse and repeated the process. In 30 minutes they brushed with Crest. They repeated this routine before bed. This routine was repeated daily for 4 weeks.
  Interventions: Biological: Tartarase
- Tartarase tray (Experimental): In the morning this group brushed with Tartarase for 30 seconds, filled a dental tray with Tartarase and applied it to the 6 lower front teeth and left it for 30 minutes, spit but did not rinse then brushed with Tartarase for another 30 seconds, spit, but did not rinse. In 30 minutes they brushed with Crest. Before bed they brushed with Crest alone. This routine was repeated daily for 4 weeks.
  Interventions: Biological: Tartarase

INTERVENTIONS:
Biological: Tartarase — Brushing with a formulation containing DNase 1 and chymotrypsin to assess its efficacy at removing accumulated calculus

SUMMARY:
This study was designed to find our whether a novel toothpaste containing safe digestive enzymes (Tartarase) was able to remove pre-existing dental tartar when compared to a well-known toothpaste (Crest). A group of 40 test subjects that had at lease 9 mm of tartar on the tongue side of the 6 lower front teeth, were randomly divided into 3 groups unknown to the the team overseeing the measurements. All the groups brushed with a toothbrush approved by the American Dental Association. Group A (20 subject) was the control group. They brushed in the morning and before bed with Crest for 2 minutes. Group B (10 subjects) brushed in the morning and before bed using the same procedure, first with Tartarase for 30 seconds, spit, but did not rinse, then repeated. After 30 minutes then brushed with Crest. Group C (10 subjects) brushed for 30 seconds with Tartarase, spit but did not rinse, then filled a dental tray with Tartarase and covered the 6 lower front teeth and waited 30 minutes, spit but did not rinse and brushed for ann additional 30 seconds with Tartarase. After 30 minutes they brushed with Crest. They brushed with crest before bed, without another Tartarase treatment. The study was a 4-week study, with tartar measured at the start (baseline), again after 2 weeks and again at the final study point of 4 weeks.

If any of the study subjects experienced anything unpleasant, they were to inform the team overseeing the study. The tartar measurements were compiled into the 3 groups and statistically analyzed to determine if there were any changes in the amount of tartar within the groups and between the groups.

DETAILED DESCRIPTION:
Quality assurance All raw data (Case Report Forms) were screened for quality assurance by the Investigators' Quality Assurance officer (QA) and found to be in compliance with protocol requirements before being sent to the Sponsor.

Data checks Not applicable Source data verification Not applicable Data dictionary

The Volpe-Manhold Index (V-MI) measures, in millimeters, calculus present on the lingual surfaces of the lower six anterior teeth. The measurement from the most inferior border of visible calculus obtained in three planes:

1. Bisecting the center of the lingual surface;
2. Diagonally through the mesial-incisal point angle of the tooth through the area of greatest calculus height; and
3. Diagonally through the distal point angle of the tooth through the area of greatest calculus height.

The primary outcome was calculus using the V-MI, all other variables are considered secondary. The calculus scores are summed to provide a total score at each clinical examination. The primary time points were at the baseline and at the after 4 weeks of product use.

Standard operating procedures Patient recruitment Subjects were recruited from site's database. Data collection During the course of the trial, the clinical site allowed monitoring by the Sponsor to check compliance with Protocol, regulations and guidelines, adequacy of the equipment and facilities, and satisfactory data collection.

Data Management Data was transferred from the case report forms (scoring charts) and entered into a database (Excel Spreadsheet) for analysis. The data was tabulated according to clinical scoring index and examination using a spreadsheet program.

Case Report Forms, questionnaires, and Subjects Diaries were entered into spreadsheets at the research site after source data verification and resolution of monitoring queries. The spreadsheets were electronically delivered to research site subcontractor for data analysis.

Data was entered using a double entry method and controlled by periodic and random validation check programming. Immediately following data validation, a data transfer was conducted to prevent modification to the spreadsheets.

Data Analysis A safety analysis set was conducted, including all subjects using the experimental gel at least a single time. A Performance analysis set consisted of all subjects providing at least one post treatment performance measurement. Only observed data was used; missing data was not imputed.

STATISTICAL ANALYSIS Subject Disposition The safety analysis set was used for describing subject disposition. Subject disposition was tabulated; the number of enrolled, exposed, prematurely terminated and completed subjects were summarized. A list of dropouts/terminations was prepared including reason for discontinuation, and time of discontinuation.

Safety Analyses Safety analyses was descriptive in nature, with SAE's and AEs tabulated by body system, preferred term, severity and relation to investigational gel. Where relevant, events were related to remote log file data. In addition, safety complaints, as described by the subjects were described and investigated.

Performance Analyses Efficacy was determined by reduction of dental calculus within treatment groups (longitudinal analysis) and between groups as compared to the control group following 4 weeks of treatment.

The primary outcome was calculus using the V-MI, as described in the Data Dictionary.

Statistical significance of mean data for age and scoring index was determined parametrically by analysis of variance for testing of differences between the product groups. Intergroup comparisons for each parameter were made by means of multiple range tests with compensation for gender, if necessary. Data from all subjects who completed the final assessment were used in the analysis.

The data for each scoring index was also analyzed by analysis of covariance using the baseline data as the covariate. The covariate (baseline data) was included in the statistics model for increased precision in determining the effect of the test products on the scores. The adjusted means generated by this procedure compensate for any variations between treatment groups that existed in the baseline data.

Longitudinal (i.e., within-treatment) comparisons were performed for V-MI means using a one-sample t-test on the changes from baseline to the final examination.

All comparisons were tested at an overall 0.05 level of significance using 2-sided tests. Summary statistics were provided at all timepoints. Safety data was summarized. Adverse events experienced by all subjects receiving test products were included in the safety analyses. All cases were checked for compliance with the study protocol, and for accuracy and completeness. Those cases which did not meet these requirements were excluded from primary analyses.

Post-power analyses for those endpoints that were determined to not be statistically significant were undertaken. Thus, sample sizes needed for a properly powered study were determined.

All adverse events reported were listed, documenting course, outcome, severity, and possible relationship to study products. Comparisons among the treatment groups were made by tabulating the frequency of subjects with one or more adverse events during the trial. If required, likelihood ratio chi square tests were used to compare the frequency of subjects experiencing adverse events among treatment groups.

Reporting for adverse events A subject may have discontinued the trial at any time for any reason. The investigator could have withdrawn a subject if, in his judgment, it was in the best interest of the subject, if the subject could not comply with the protocol, or if a Serious Adverse Event occurred. If a subject withdrew, the reason was recorded in the CRF End of Study Statement and signed by the Investigator.

Risk Assessment Risk is the product of the likelihood that an adverse medical event will occur, times the severity of the event. A comprehensive Risk Analysis was conducted for the Tartarase gel to indicate it was safe for human use. The risk analysis report was available upon request.

Adverse Events Definitions An Adverse Event (AE) is any untoward medical occurrence (sign, symptom, illness, abnormal laboratory value, or other medical event) in a subject. This definition does not imply that there is a relationship between the adverse event and the device under investigation. (Significant device failure may constitute an adverse event if an undesirable experience occurs).

An Adverse Device Effect (ADE) is any untoward and unanticipated response to a medical device. This definition includes any event resulting from insufficiencies or inadequacies in the instructions for use or the deployment of the device, or any event that is a result of a user error.

Serious Adverse Event (SAE)

A serious adverse event (SAE) is any adverse event that:

Led to death Led to a serious deterioration in the health of the subject that resulted in a life-threatening illness or injury Resulted in a permanent impairment of a body structure or a body function Required in-subject hospitalization or prolongation of existing hospitalization Resulted in medical or surgical intervention to prevent permanent impairment to body structure or a body function Led to fatal distress, a congenital abnormality, birth defect or death An unanticipated adverse event is any serious, study product related adverse event, if that event was not previously identified in the risk analysis and informed consent form in nature, severity, or frequency.

Adverse events are graded according to severity as follows: Mild: Sign or symptom, usually transient, requiring no special treatment and generally not interfering with usual activities. Moderate: Sign or symptom, which may be ameliorated by simple therapeutic measures; yet, may interfere with usual activity. Severe: Sign or symptom that are intense or debilitating and that interfere with usual activities. Recovery is usually aided by therapeutic measures.

The Investigator reported all Adverse Events which occurred with each subject throughout the study and follow-up period and recorded them in the CRF Adverse Events Investigation Form. The Investigator categorized Adverse Events according to:

Serious or non-serious Severity Anticipated or unanticipated Relationship to device use INVESTIGATOR REPORTING OF AES

The Investigator would have reported all serious adverse events (SAEs) to Pontis Biologics by telephone as soon as becoming aware of them. A written follow-up report would have been emailed or faxed to Pontic Biologics and the reviewing IRB within 24 hours and would have included the following information:

Nature of SAE Statement regarding the degree to which it is considered device related, and rationale Results of any diagnostic tests that were performed Description of any treatment implemented Statement of subject's current clinical status Investigator's signature and date

Non-serious adverse events that were unanticipated and may have been study product related were reported to the Pontic Biologics by telephone within 24 hours. A written follow-up report was emailed or faxed to Pontis Biologics within 5 working days and included the following information:

Nature of adverse effect (AE) Statement as to why it is considered unanticipated Statement as to the degree to which it is considered device related, and rationale Results of any diagnostic tests that were performed Description of any treatment implemented Statement of subject's current clinical status Change Management Not applicable Sample size assessment See statistical analysis Plan for missing data Not applicable Statistical Analysis The primary outcome was calculus using the V-MI, and all other variables are considered secondary. Statistical significance of mean data for age and scoring index was determined parametrically by analysis of variance for testing of differences between the product groups. Intergroup comparisons for each parameter were made by means of multiple range tests with compensation for gender, if necessary. Data from all subjects who completed the final assessment were used in the analysis.

The data for each scoring index was also analyzed by analysis of covariance using the baseline data as the covariate. The covariate (baseline data) was included in the statistics model for increased precision in determining the effect of the test products on the scores. The adjusted means generated by this procedure compensate for any variations between treatment groups that existed in the baseline data.

Longitudinal (i.e., within-treatment) comparisons were performed for V-MI means using a one-sample t-test on the changes from baseline to the final examination.

All comparisons were tested at an overall 0.05 level of significance using 2-sided tests. Summary statistics were provided at all timepoints. Safety data was summarized. Adverse events experienced by all subjects receiving test products were included in the safety analyses. All cases were checked for compliance with the study protocol, and for accuracy and completeness. Those cases which did not meet these requirements were excluded from primary analyses.

Post-power analyses for those endpoints that were determined to not be statistically significant were undertaken. Thus, sample sizes needed for a properly powered study were determined.

All adverse events reported were listed, documenting course, outcome, severity, and possible relationship to study products. Comparisons among the treatment groups were made by tabulating the frequency of subjects with one or more adverse events during the trial. If required, likelihood ratio chi square tests were used to compare the frequency of subjects experiencing adverse events among treatment groups.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study, each subject must have:

1. Provided written informed consent to participate in the study;
2. Adult subjects aged 18 years and older, that were in good health;
3. Agreed not to participate in any other oral/dental product studies during the course of this study and used only the assigned oral hygiene products during the entire study (including toothbrushes, toothpastes, home remedies, floss or other products like chewing gum, mouthwashes, tongue cleaners, etc.);
4. Agreed to refrain from the use of any elective dentistry (including a non-study dental prophylaxis) until the study had been completed;
5. Agreed to refrain from the use of any non-study oral hygiene and whitening products;
6. Been in good general health, as determined by the investigator/designee based on a review of the health history/update for participation in the study;
7. Had six mandibular anterior teeth with no crowns or veneers;
8. Agreed to comply with the study procedures and schedule, including the follow up visits;
9. Had at least 9mm of dental calculus on the mandibular anterior six teeth and reported that they had received a dental cleaning in previous 2-6 months.
10. Healthy Volunteers

Exclusion Criteria:

1. Had a medical condition requiring antibiotic premedication prior to dental procedures;
2. Regularly used chlorhexidine mouth rinse;
3. Had any oral condition or pathosis that could interfere with study compliance and/or examination procedures (e.g., widespread caries, chronic neglect, advanced periodontal disease);
4. Had current or history of oral cavity cancer or oropharyngeal cancer;
5. Were pregnant or nursing by subject report;
6. Did not brush regularly;
7. Had any condition that might have made it unsafe for the subject to participate in this study, at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Tartarase Efficacy | 4 weeks
  Assess the change in calculus abundance measured by the V-MI in groups brushing with Crest, the Tartarase brushing group and the Tartarase tray group.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Mynarcik, PhD, Study Chair — Pontis Biologics, Inc.
Locations (1):
- Pontis Biologics, Inc, Huntington, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] VOLPE AR, MANHOLD JH, HAZEN SP. IN VIVO CALCULUS ASSESSMENT. I. A METHOD AND ITS EXAMINER REPRODUCIBILITY. J Periodontol (1930). 1965 Jul-Aug;36:292-8. doi: 10.1902/jop.1965.36.4.292. No abstract available. PMID 14326695
- [Derived] Milleman KR, Deener G, Milleman JL, Mish B, Schuller R, Mynarcik D. A proof of principle investigation of a novel enzyme formulation on dental calculus deposition: a 4-week randomized human clinical trial. BMC Oral Health. 2024 Jun 22;24(1):720. doi: 10.1186/s12903-024-04498-x. PMID 38909189